CLINICAL TRIAL: NCT04808674
Title: EvalUation of REmediation Programs for Patients Suffering From Mild Cognitive Deficits After CAncer
Brief Title: Remediation for Mild Cognitive Deficits After Cancer
Acronym: EURECA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_1018; 2021-A00798-33 (Other: ID-RCB)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Remediation; Breast Cancer
Keywords: Neuropsychology; psychological distress; quality of life; rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based cognitive remediation program (Experimental): Patients are admitted to the day hospital 2 days a week for 6 weeks and participate in a group-based (4 patients per group) rehabilitation program conducted by a multidisciplinary team including a PMR doctor, a neuropsychologist, an occupational therapist, and a physical activity monitor).
  Interventions: Behavioral: Cognitive remediation program
- One-on-one cognitive remediation program (Experimental): Patients are admitted to the day hospital 5 days a week for 6 weeks and participate in a one-on-one intensive rehabilitation program conducted by a multidisciplinary team including a speech therapist, neuropsychologist, occupational therapist, physiotherapist, physical activity monitor and a psychologist.
  Interventions: Behavioral: Cognitive remediation program

INTERVENTIONS:
Behavioral: Cognitive remediation program — Evaluation of REmediation programs for patients suffering from mild cognitive deficits after Cancer

SUMMARY:
Cancer survival rates have improved significantly over the past decades and patients now experience a number of side effects including cancer-related cognitive impairment (CRCI): problems with memory, executive function, attention, and difficulties performing two tasks at the same time. The frequency of CRCI in cancer patients is estimated to be between 10 to 40%, and more than 50% of patients describe difficulties in their daily life. These cognitive difficulties negatively impact the patient's quality of life as well as that of their family, and can also have negative consequences for their social and professional reintegration once cancer treatment is finished. Despite an increasing number of studies on CRCI, a standard of care for patients with CRCI after breast cancer is yet to be established. In the absence of clear directives, and in an attempt to respond to the increasing demand to provide care for breast cancer patients with CRCI, physical medicine and rehabilitation units in France have started providing day-hospital multidisciplinary interventions. The objective of this project is to use the single case experimental design method to investigate the efficacy of two such rehabilitation programs: a group-based program and a one-on-one program.

ELIGIBILITY:
Inclusion Criteria:

* Treated in the past for breast cancer with chemotherapy, surgery, and / or radiotherapy,
* Admitted as a day patient at the Henry Gabrielle Hospital or the Pontchaillou CHU Hospital during the study,
* Given free, informed consent in writing after being informed orally and in writing of the how the study will proceed.

Exclusion Criteria:

* Presence of another active cancer,
* Ongoing chemotherapy and/or radiotherapy treatment,
* Active progression of breast cancer,
* History of neurological or psychiatric conditions,
* Major disturbances in comprehension that prevent them giving free, informed consent,
* Pregnant, parturient or breastfeeding women,
* Person under a legal protection measure such as guardianship or curatorship,
* People not affiliated to a social security scheme (French Social Security) or beneficiaries of a similar scheme.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
Self-reported cognitive function | 16 weeks
  The Fact-COG questionnaire assesses subjective cognitive impairment. The score directly reflects the patient's feelings about/perceptions of their cognitive function over the previous week. A total score out of 132 is obtained as well as 4 subscales: Perceived Cognitive Impairments (0-72), Impact on Quality of Life (0-16), Comments from Others (0-16), and Perceived Cognitive Abilities (0-28).

SECONDARY OUTCOMES:
Neuropsychological function | 16 weeks
  Neuropsychological function will be measured using three sub-tests of the Test of Attentional Performance (alertness, covert shift of attention, divided attention), the Paced Auditory Serial Addition Test, the Montreal Cognitive neuropsychological Assessment, and the Symbol Digit Modalities Test.
Psychological distress | 16 weeks
  Psychological distress will be measured using 4 questionnaires: The Hospital Anxiety and Depression Scale; the Brief Symptom Inventory-18; the Rosenberg self-esteem scale; the MCQ-30 Meta-cognition self-report questionnaire.
Quality of Life with FACT-B questionnaire | 16 weeks
  The FACT-B questionnaire assesses cancer-related quality of life. A total score out of 148 is obtained as well as 5 subscales: Physical Well-Being (0-28), Social/Family Well-Being (0-28), Functional-Well-Being (0-28), Emotional Well-Being (0-24), and Breast Cancer Subscale (0-40).
Fatigue | 16 weeks
  The FACTIT-Fatigue questionnaire assesses fatigue/ tiredness and its impact on daily activities and functioning in chronic disease. A total score out of 52 is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JACQUIN-COURTOIS, PhD, Principal Investigator — Service de médecine physique et de réadaptation, HCL,
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Groupement hospitalier sud - Hôpital Henry Gabrielle - Service de médecine physique et de réadaptation, Lyon
  - Hôpital Pontchaillou - Service de Médecine Physique et de Réadaptation, Rennes